CLINICAL TRIAL: NCT02606019
Title: The Use of Biomarkers in Predicting Dengue Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiti Tunku Abdul Rahman (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Gary Kim Kuan Low, Dr., Universiti Tunku Abdul Rahman
Other Study IDs: NMRR-15-1045-25937
Record Dates: First submitted 2015-11-09; First posted 2015-11-17 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Dengue
Keywords: Pentraxin 3; Vascular Endothelial Growth Factor; dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum/plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The burden of dengue infection has increased due to the current non-specific classification. A pilot study was conducted to evaluate the five of the biomarkers: neopterin, vascular endothelial growth factor (VEGF), thrombomodulin, Vascular Cell Adhesion Molecule 1 (VCAM-1) and pentraxin 3 (PTX-3). VEGF and PTX-3 was the only two potential biomarkers in differentiating severe dengue from non-severe dengue cases. The analysis between severe dengue and non-severe dengue cases indicated that only VEGF was able to discriminate the two categories. Though VCAM-1 and PTX-3 were not statistically significant, the p-values were at the margin of the pre-determined p-value of less than 0.05.

Hence, this study aims to evaluate VEGF and PTX-3 levels in differentiating severe dengue from non-severe dengue cases. The secondary objective is to evaluate the correlation of VEGF and PTX-3 levels with full blood count (platelet, white blood cell count and haematocrit) and liver function test (alanine aminotransferase and aspartate).

DETAILED DESCRIPTION:
The burden of dengue infection has increased due to the current non-specific classification. A pilot study was conducted to evaluate the five of the biomarkers: neopterin, vascular endothelial growth factor (VEGF), thrombomodulin, Vascular Cell Adhesion Molecule 1 (VCAM-1) and pentraxin 3 (PTX-3). VEGF and PTX-3 was the only two potential biomarkers in differentiating severe dengue from non-severe dengue cases. The analysis between severe dengue and non-severe dengue cases indicated that only VEGF was able to discriminate the two categories. Though VCAM-1 and PTX-3 were not statistically significant, the p-values were at the margin of the pre-determined p-value of less than 0.05.

Hence, this study aims to evaluate VEGF and PTX-3 levels in differentiating severe dengue from non-severe dengue cases. The secondary objective is to evaluate the correlation of VEGF and PTX-3 levels with full blood count (platelet, white blood cell count and haematocrit) and liver function test (alanine aminotransferase and aspartate).

This is a prospective cohort study in which the patient will be followed up from the day of presentation to the attending practitioner until the patient is discharged. The blood samples will be obtained daily during the follow-up. The demography and clinical final diagnosis will be obtained from the medical record of the patient.

This study will aid triaging of dengue cases thereby reducing the need of unnecessary admission and better focused management to those might develop complication of dengue infection. This in turn reduces the workload and cost of the treating the dengue infection.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are age 15 or more.
* Participants must be recruited within the first three days of fever.
* Positive dengue by NS1Ag. Confirmed later on by paired dengue IgM/IgG.
* Final diagnosis of severe dengue or non-severe dengue.

Exclusion Criteria:

* Participants who are less than 15 years old.
* Pregnant mothers.
* Participants should not have autoimmune disorder, haematological disorder, cancer, cardiovascular disease, on long term warfarin and aspirin.
* Participants who have been previously treated with dengue infection (secondary dengue infection will be excluded by dengue IgM/IgG).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients will be recruited from primary care and followed up in the hospital if they were admitted.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (%) of biomarkers (PTX3 and VEGF) | upon study completion, 3 years
  The measures will be analysed using Receiver Operating Characteristics (ROC) during the first 4 days of illness to predict the outcome of dengue infection (severe dengue versus non-severe dengue. Both univariate and multivariate analysis will be performed to identify and control for confounding factors.
Specificity (%) of biomarkers (PTX3 and VEGF) | upon study completion, 3 years
  The measures will be analysed using Receiver Operating Characteristics (ROC) during the first 4 days of illness to predict the outcome of dengue infection (severe dengue versus non-severe dengue. Both univariate and multivariate analysis will be performed to identify and control for confounding factors.
Positive predictive value (%) of biomarkers (PTX3 and VEGF) | upon study completion, 3 years
  The measures will be analysed using Receiver Operating Characteristics (ROC) during the first 4 days of illness to predict the outcome of dengue infection (severe dengue versus non-severe dengue. Both univariate and multivariate analysis will be performed to identify and control for confounding factors.
Negative predictive value (%) of biomarkers (PTX3 and VEGF) | upon study completion, 3 years
  The measures will be analysed using Receiver Operating Characteristics (ROC) during the first 4 days of illness to predict the outcome of dengue infection (severe dengue versus non-severe dengue. Both univariate and multivariate analysis will be performed to identify and control for confounding factors.

SECONDARY OUTCOMES:
Correlation of routine blood parameters with PTX 3 and VEGF. | upon study completion, 3 years
  Pearson's/Spearmann correlation routine blood parameters (ALT, AST, PLT count, HCT and WBC count) with the biomarkers to identify possible prognostic value.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Low, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (2):
- Malaysia (2):
  - Ampang Hospital, Ampang, Selangor
  - Klinik Kesihatan Ampang (Ampang Health Clinic), Ampang, Selangor